CLINICAL TRIAL: NCT03163836
Title: Impact of Concomitant Surgical Atrial Fibrillation Ablation in Patients Undergoing Double Valve Replacement
Brief Title: Concomitant Surgical Atrial Fibrillation Ablation in Double Valve Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Weida Zhang, Director of Cardiovascular Surgery, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: RS2016003
Record Dates: First submitted 2017-04-03; First posted 2017-05-23 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Valvular Heart Disease
Keywords: Double Valve Replacement; Atrial Fibrillation Ablation
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- double valve replacement group: Patients received aortic+mitral valve replacement at Guangzhou General Hospital of Guangzhou Military Command with persistent or long-standing atrial fibrillation(AF) but did not received concomitant AF ablation. Persistent AF was defined as AF lasting more than 7 days and long-standing persistent AF as continuous AF for more than 12 months. Exclusion criteria for consideration for concomitant AF ablation includes >70 years old, left atrium (LA) diameter >7 cm, or preoperative left ventricle (LV) ejection fraction < 40% and patients falls in these criteria were excluded from this group.
  Interventions: Procedure: double valve replacement
- surgical ablation group: Patients received aortic+mitral valve replacement at Guangzhou General Hospital of Guangzhou Military Command with persistent or long-standing atrial fibrillation(AF) and received concomitant surgical ablation. Persistent AF was defined as AF lasting more than 7 days and long-standing persistent AF as continuous AF for more than 12 months.
  Interventions: Procedure: double valve replacement; Procedure: surgical ablation

INTERVENTIONS:
Procedure: double valve replacement — After median sternotomy, cardiopulmonary bypass was established via bicaval and aortic cannulation. After cross-clamping of the aorta and cardioplegia, mitral and aortic replacement were performed. Supplementary procedures such tricuspid annuloplasty, ascending aorta replacement and coronary artery bypass grafting were performed as required. The left atrial appendage was excised to avoid thrombus formation.
  Other Names: tricuspid annuloplasty; ascending aorta replacement; coronary artery bypass grafting
Procedure: surgical ablation — Both left and right atrial ablation were performed using a bi-polar radiofrequency ablation clamp.
  Other Names: tricuspid annuloplasty; ascending aorta replacement; coronary artery bypass grafting
  Groups: surgical ablation group

SUMMARY:
Current European Society of Cardiology Guidelines recommend concomitant atrial fibrillation (AF) ablation for all symptomatic patients undergoing other cardiac surgeries, but the safety and potential benefits of concomitant atrial fibrillation (AF) ablation at the time of double valve replacement remains unexamined. A retrospective review of patients with AF who underwent double valve replacement with or without concomitant surgical ablation in our institute starting from April 2006.

DETAILED DESCRIPTION:
Persistent AF was defined as AF lasting more than 7 days and long-standing persistent AF as continuous AF for more than 12 months. Concomitant surgical AF ablation was offered to suitable patients as determined by the surgeon, and patients then decided whether to undergo the additional procedure.

The operations were performed through median sternotomy and under cardiopulmonary bypass. The bipolar ablation clamp was positioned precisely around the pulmonary veins (PV) for bilateral circular ablation. After Marsh ligament cutting and cross-clamping the ascending aorta, the left atrial appendage was resected and left atrial cavity exposed through an incision behind the interatrial groove. Then, linear ablations were performed between the left and right inferior PVs, between the left and right superior PVs, between the left superior PV and the opening of the left atrial appendage, and between the line connecting bilateral inferior PVs and the mitral valve isthmus. Ablation at the right atrium was then performed. Briefly, the bipolar ablation clamp was positioned around the inferior vena cava (IVC) and right atrial appendage for circular ablation. An L-shaped incision was then made on the anterior wall of the right atrium and linear ablations were performed vertically from the incision to the interatrial groove and tricuspid annulus, to the ablation ring around the right atrial appendage, and from the superior vena cava to the ablation ring around the inferior vena cava.

The left atrial appendage was always excluded by resection and the incision was closed with continuous running stitches. Temporary pacemakers were placed in all patients and activated when heart rate was less than 70 beats per minute.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to our institute with valvular heart disease requiring double valve replacement and also present with persistent or long-standing persistent atrial fibrillation.
* Persistent AF was defined as AF lasting more than 7 days and long-standing persistent AF as continuous AF for more than 12 months. First cardiac surgery, age<70 years. left atrium diameter measured by transthoracic echocardiography<7cm. Left ventricular ejection fraction > 40%

Exclusion Criteria:

* >70 years old, with LA diameter >7 cm, or with LV ejection fraction < 40% , repeated cardiac surgery, concomitant tricuspid valve replacement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented to our institute with valvular heart disease requiring double valve replacment and also present with persistent or long-standing persistent atrial fibrillation. Persistent AF was defined as AF lasting more than 7 days and long-standing persistent AF as continuous AF for more than 12 months
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-04-01 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
mortality | from the date of the surgery until the date of death, assess up to 120 months
  mortality from any cause
sinus rhythm rate | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  sinus rhythm rate examined by 24h holter monitoring
stroke | from the date of surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  perioperative stroke
third degree heart block requiring permanent pacemaker implantation | from the date of surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  third degree heart block diagnosed via ECG

SECONDARY OUTCOMES:
perioperative morbidities | from the date of surgery until the date of first documented progression or date of death from any cause, assess up to 30 days
  Redo for bleeding; Low cardiac output syndrome; Renal failure requiring dialysis; Pneumonia;
Warfarin-related bleeding | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  bleeding events occurred during the period when warfarin was used
Thromboembolic events | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  thromboembolic events
New York Heart Function classification | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  New York Heart Function classification
warfarin requirement | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  oral warfarin requirement over 6 moths after the surgery
left ventricular ejection fraction | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  left ventricular ejection fraction measured by transthoracic echocardiography
left atrium diameter | from 6 months after surgery until the date of first documented progression or date of death from any cause, assess up to 120 months
  left atrium diameter measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Weida Zhang, MD, Principal Investigator — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided